CLINICAL TRIAL: NCT06124144
Title: Safety and Pharmacokinetics of Oleylphosphocholine (OlPC), Administered Orally in Healthy Adults: A Phase 1, Single Center, Open-label, Staggered, Dose-escalation Trial
Brief Title: Safety and Drug Absorption of Orally Administered Oleylphosphocholine (OlPC) in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The risk-benefit ratio changed
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TT4CL_EKUT; 2021-004936-27 (EudraCT Number)
Record Dates: First submitted 2023-08-31; First posted 2023-11-09 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-06

CONDITIONS: Leishmaniasis
MeSH Terms: conditions — Leishmaniasis | interventions — oleylphosphocholine

STUDY DESIGN:
Intervention Model Description: 3+3 design for ascending doses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oleylphosphocholine capsules (IMP) oral administration (Experimental): Participants will receive once Oleylphosphocholine (capsule/s) orally as a single dose under fed conditions.
  Interventions: Drug: Oleylphosphocholine

INTERVENTIONS:
Drug: Oleylphosphocholine — The trial is a dose escalation trial that follows a 3+3 approach. The sample size is determined by a decision-making algorithm and by the tolerability of the study drug in the study participants. This design follows predetermined rules that help identify notable toxicities in time with a reasonable degree of accuracy. The initial dose will be 50mg OlPC (1 capsule) and participants in subsequent cohorts will receive 100mg (2 capsules), 150mg (3 capsules), 200mg (4 capsules), 250mg (5 capsules), or 300mg (6 capsules) if the previous doses are tolerated. The study ends when the last cohort is completed or when it is determined that a dose (within a cohort) is not tolerable.
  Other Names: OlPC

SUMMARY:
The goal of this interventional study is to assess the safety and tolerability of OlPC and to characterize the pharmacokinetics (PK) of OlPC following single, ascending doses administered orally in healthy-fed subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females of non-childbearing (see below) potential.

   1. 18 - 60 years of age.
   2. BMI between 20-30 and body weight from 55-100 kg.
2. Females of non-childbearing potential defined as follows:

   1. Surgically sterile (history of bilateral tubal ligation/occlusion, bilateral oophorectomy or hysterectomy) or
   2. Postmenopausal, defined as amenorrhea for ≥ 12 consecutive months prior to screening without an alternative medical cause. A follicle-stimulating hormone (FSH) level will be measured to confirm postmenopausal status.
3. Males must agree:

   1. to use a latex condom during any sexual contact with while participating in the study and for 3 months following discontinuation from this study, even if he has undergone a successful vasectomy.
   2. to refrain from donating semen or sperm during study participation and for 3 months after discontinuation from this study.
4. Able and willing (in the investigator's opinion) to comply with all trial requirements.
5. Available to participate in follow-up for the duration of trial.
6. Living in the area close enough to be able to attend all follow-up visits.
7. General good health based on the definition in BreithauptGrögler et al. 2017 and based on history, clinical examination and laboratory results.
8. Signed informed consent.
9. Consent to provide clinical history and if necessary consent that the study team is allowed to contact the family doctor of the participant.
10. All subjects are forbidden from donating blood while on study drug and for 3 months after discontinuation from this study

Exclusion Criteria:

1. Any confirmed or suspected immunosuppressive or immunodeficient state, asplenia, recurrent, severe infections and chronic immunosuppressant medication (more than 14 days) within the past 6 months.
2. Any history of or signs of hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, or neurologic clinical significant abnormalities.
3. History of chronic infections (e.g., hepatitis В or С) and chronic inflammation.
4. History of significant, acute or chronic gastrointestinal, hepatic, cardiac or renal disorders.
5. History of leishmaniasis.
6. History of hypersensitivity to the excipients present in the investigational medicinal product or to any drug with similar chemical structure (Miltefosine).
7. Use of immunoglobulins or blood products within 3 months prior to enrolment.
8. Receipt of any investigational medicinal product in the 30 days preceding enrolment, or planned receipt during the trial period.
9. Participation in other clinical trials or observation period of competing trials.
10. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ in the last five years).
11. Mental disorders or other psychiatric conditions (including depression).
12. The average alcohol intake greater than 24 g pure alcohol per day for men or greater than 12 g pure alcohol per day for women (including history of possible addiction) and alcohol consumption on more than five days a week.
13. Suspected or known injecting drug abuse in the 5 years preceding enrolment.
14. Participants unable to be closely followed for social, geographic or psychological reasons.
15. Any clinically significant abnormal finding on biochemistry or hematology blood tests, urine analysis or clinical examination.
16. History of seizure, except for sporadic childhood febrile convulsions.
17. Sjoegren-Larsson-Syndrome (SLS).
18. Participants who are unwilling to ingest the food provided.
19. Any other significant disease, disorder or finding which, in the opinion of the investigator, may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Subject incidence of treatment-emergent adverse events at administration and follow-up visits | Participants are followed up for 21 days and an additional telephone visit 35 days after drug administration will be conducted before dismissing the participant.

SECONDARY OUTCOMES:
Cmax | 21 days
  Maximum observed concentration in plasma after single dose (µg/mL)
Tmax | 21 days
  Time of maximum observed concentration (h)
AUC0-t | 21 days
  Area under the curve (AUC) from time 0 to the time of the last measurable concentration, calculated using the Linear Up / Log Down trapezoidal rule (h*µg/mL)
AUC0-24 | 21 days
  Area under the curve from time 0 to hour 24 (single-dose only), calculated using the Linear Up / Log Down trapezoidal rule (h*µg/mL)
AUC0-inf | 21 days
  Area under the curve from time 0 to infinity (single-dose only), calculated as AUC0-inf = AUC0-t + Ct / λz, where Ct is the last observed quantifiable concentration and λz is the elimination rate constant (h*µg/mL)
t1/2 | 21 days
  Elimination half-life, calculated as ln(2) / λz (h)
AUCres | 21 days
  Residual Area: extrapolated area (single-dose) calculated as AUCres = 100 (AUC(0-inf) - AUC(0-t)) / AUC(0-inf)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Tropical Medicine, Tübingen, Germany

REFERENCES:
- See also: Official website — https://tt4cl-h2020.eu/